CLINICAL TRIAL: NCT05718076
Title: A Prospective, Observational Study to Investigate Visual Outcome After Trifocal Intraocular Lens Implantation in High Myopic Patient With Different Meta-PM Grading Fundus Appearance.
Brief Title: Trifocal Intraocular Lens in High Myopic Patients With Different Meta-PM Grading
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: SHAIER2021IRB04-1
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Myopia; Intraocular Lens Complication
MeSH Terms: conditions — Myopia | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: Eyes are categorized by fundus META-PM as grade 0
  Interventions: Procedure: cataract surgery
- group 2: Eyes are categorized by fundus META-PM as grade 1
  Interventions: Procedure: cataract surgery
- group 3: Eyes are categorized by fundus META-PM as grade 2
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — Phacoemulsification combined trifocal lens implantation
  Other Names: Phacoemulsification combined trifocal lens implantation

SUMMARY:
Study the postoperative visual quality and safety of trifocal intraocular lenses implanted in patients with different levels of myopic maculopathy stages according to Meta-PM staging (stage 0-2).

DETAILED DESCRIPTION:
Cataracts occur in patients with high myopia who are younger than age related cataract patients. These relatively young cataract patients have a higher demand for lens removal, and therefore have a higher acceptance of multifocal intraocular lenses. Some current studies have shown that the implantation of multifocal intraocular lenses in patients with high myopia has achieved good visual effects after surgery. As we all know, high myopia is associated with a higher incidence of postoperative complications, and high myopia macular degeneration can affect postoperative visual effects and patient satisfaction. However, there is no research to evaluate the clinical effect of multifocal intraocular lens implantation in patients with high myopia according to different fundus Meta-PM classifications.Therefore, the purpose of this study is to study the postoperative visual quality and safety of trifocal intraocular lenses implanted in patients with different levels of myopic maculopathy stages according to Meta-PM staging (stage 0-2).

ELIGIBILITY:
Inclusion Criteria:

Age-related cataract 26mm ≤ AL ≤ 30mm Pre-op corneal astigmatism ≤ 1.0 D (IOLMaster 700, Carl Zeiss Meditec AG); Eyes with angle kappa ≤ 0.50 mm (iTrace); Eyes with corneal spherical aberration ≤ 0.30 (iTrace); High order aberration ≤ 0.3 (iTrace). 2.2 ≤ pupil size ≤ 5.5mm Meta-PM classification grade 0, 1 and grade 2 with low risk of MM progression No maculopathy(complete and continuous macular retinal structure revealed by OCT)

Exclusion Criteria:

Combined with Glaucoma, serious fundus pathological change, intracranial tumor Any systemic disease may cause secondary vision impair Synechia Other ocular surgery history history of serious cardiopulmonary or cerebrovascular diseases, and serious mental and psychological diseases Sensitive, anxiety perfectionist Any myopic macular lesion, Posterior staphyloma, any Plus lesions in meta-PM classification, including but not limited to CNV, lacquer cracks, dome-shaped macula, Fuchs spot, etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who plan to have cataract surgery in the near future
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 12 months
  Monocular BCVA, UCVA(5m), BCIVA, UIVA(60cm) and BCNVA, UNVA(40cm) VA

CONTACTS AND LOCATIONS:
Overall Officials: Hua Fan, Principal Investigator — Shanghai Aier Eye Hospital
Locations (2):
- China (2):
  - Hua Fan, Shanghai
  - Shanghai Aier Eye Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No